CLINICAL TRIAL: NCT00082134
Title: A Phase II Study of ILX651 Administered Intravenously Daily for Five Consecutive Days Every 21 Days in Patients With Hormone-Refractory Prostate Cancer Previously Treated With Docetaxel
Brief Title: Study of ILX651 in Patients With Hormone-Refractory Prostate Cancer Previously Treated With Docetaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILX651-241
Record Dates: First submitted 2004-04-29; First posted 2004-05-04 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Hormone-refractory Prostate Cancer
Keywords: Prostate cancer; Hormone-refractory prostate cancer; HRPC; Prostate; Docetaxel; PSA progression; PSA progressed
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tasidotin

INTERVENTIONS:
Drug: ILX651

SUMMARY:
This is a Phase II, non-randomized, open label study of ILX651 in patients with hormone-refractory prostate cancer previously treated with docetaxel. Approximately 40 patients will be enrolled in this study that is expected to last 24 months. All patients will be treated with ILX651 administered IV daily for 5 consecutive days every 21 days. The primary objective of this study is to determine the PSA response rate. The secondary objectives are to determine response of measurable disease, duration of response, time to PSA progression, time to treatment failure, survival, safety and tolerability, and pharmacokinetic profile of ILX651.

ELIGIBILITY:
Inclusion Criteria:

* Patient has hormone-refractory prostate cancer (HRPC) as evidenced by PSA progression or progression of measurable disease.
* Patient has greater than 25% increase in 2 consecutive tests in which the first increase in PSA should occur a minimum of 1 week apart.
* Patients on androgen deprivation treatment and will continue on androgen deprivation treatment during study participation except for patients who are post orchiectomy.
* Patient has evidence of metastatic disease by positive bone scan or evidence of progressive metastatic disease by CT scan.
* Patient has been treated with at least 1 prior hormone therapy or is post orchiectomy.
* Patient has been previously treated at a minimum for an 8-week treatment period on a docetaxel-based regimen for metastatic HRPC.
* Patient has PSA at least 5 ng/mL or greater.
* Patient has testosterone less than 50 ng/dL.
* Patient ECOG performance status of 0 or 1.
* Patient has life expectancy of greater than 8 weeks.
* Patient meets lab values: A. Absolute neutrophil count at least 1,500/mm^3 or greater; B.Platelet count at least 100,000/mm^3 or greater; C. Serum creatinine at least 1.5 mg/dL or less or creatinine clearance at least 60 mL/min or greater; D. Bilirubin less than 2.0 mg/dL. E. AST and ALT less or equal to 2.5 times upper limit of normal
* Any chemotherapy, major surgery, or irradiation must be completed at least 4 weeks prior to study drug.
* Patient recovered from clinically significant toxicities from prior treatment.

Exclusion Criteria:

* Prior treatment with 2 or more prior chemotherapy regimens.
* Concurrent treatment with an estrogen-containing agent including diethylstilbestrol (DES).
* Prior flutamide (Eulexin) within past 4 weeks, prior bicalutamide (Casodex) within past 6 weeks, or prior nilutamide (Nilandron) within past 6 weeks.
* Prior strontium or samarium or other radioisotope therapy.
* Prior radiation therapy to greater than 25% of the bone marrow (e.g., no whole pelvic irradiation is allowed).
* Uncontrolled congestive heart failure or angina, patients with a history of myocardial infarction within 2 months of enrollment.
* Patients with uncontrolled hypertension.
* Pre-existing cardiac, pulmonary, neurologic or other disease that would preclude study participation.
* Documented untreated central nervous system (CNS) metastases. However, patients with treated CNS metastases that have been stable are eligible.
* Any significant concurrent disease or illness, or psychiatric disorders or alcohol or chemical abuse that would preclude study participation.
* Active secondary malignancy except non-melanoma skin cancers.
* Known, active infection, or known HIV positive or presence of an AIDS related illness.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Kansas City Cancer Centers, Lenexa, Kansas
  - Kansas City Cancer Centers, Overland Park, Kansas
  - Kansas City Cancer Centers- Central, Kansas City, Missouri
  - Cancer Center of North Carolina- Cary, Cary, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Sammons Cancer Center, Dallas, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Joe Arrington Cancer Center, Lubbock, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington